CLINICAL TRIAL: NCT02543983
Title: The Neurobiology of Suicide
Brief Title: Neurobiology of Suicide
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 150188; 15-M-0188
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Healthy Volunteers; Depression
Keywords: Neurobiology; Suicide; Ketamine; Major Depressive Disorder; Biomarkers
MeSH Terms: conditions — Depression; Suicide; Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 1 (Experimental): Ketamine Hydrochloride infusion
  Interventions: Device: Magnetic Resonance Imaging scanner, 3T; Device: NeurOptics PLRTM-3000 Pupillometer; Device: Experimental Anxiety Devices; Device: Magnetic Resonance Imaging scanner, 7T; Drug: Ketamine Hydrochloride

INTERVENTIONS:
Device: Magnetic Resonance Imaging scanner, 3T — Non-significant risk device used for brain imaging.
Device: NeurOptics PLRTM-3000 Pupillometer — The NeurOptics PLRTM-3000 Pupillometer will use quantitative infrared technology to objectively and accurately measure pupil size and dynamics.
Device: Experimental Anxiety Devices — Acoustic startle and shock devices are used to evaluate anxious responses to stimuli. Both are considered non-significant risk under this study.
Device: Magnetic Resonance Imaging scanner, 7T — Non-significant risk device used for brain imaging.
Drug: Ketamine Hydrochloride — A non-competitive N-methyl-D-aspartate receptor antagonist. This drug is exempt from FDA IND review under the study.

SUMMARY:
Background:

There are no good treatments for people considering suicide. Researchers want to study suicide with questions, blood tests, brain imaging, and sleep studies. They hope to better understand suicide, so they can help suicidal people.

Objective:

To understand what happens in the brain when someone has thought about or attempted suicide.

Eligibility:

Group 1: Adults ages 18 70 who have thought about or attempted suicide recently

Group 2: Adults ages 18 70 who have thought about or attempted suicide in the past

Group 3: Adults ages 18 70 who have depression or anxiety, but have never thought about suicide

Group 4: Healthy volunteers the same ages.

Design:

Participants will be screened in another protocol. Adults who have recently thought about or attempted suicide must be referred by a doctor. They may do up to 3 phases of this study. Groups 2, 3 and 4 will do only Phase 1 and will not get ketamine.

Phase 1: 1 week in hospital. Participants will have:

Physical exam.

Questions about thoughts and feelings.

Thinking and memory tests and simple tasks.

Blood and urine tests.

Two MRI scans. Participants will lie on a table that slides into a metal cylinder that takes pictures. They will have a coil over their head and earplugs and do a computer task.

Sleep test. Disks and bands will be placed on the body to monitor it during sleep.

Magnetic detectors on their head while they perform tasks.

A wrist monitor for activity and sleep.

Lumbar puncture (optional). A needle will collect fluid from the back.

Shock experiments (optional). Participants will observe pictures and sounds and feel a small shock on the hand.

Phase 2: 4 days in hospital. A thin plastic tube will be placed in each arm, one for blood draws, the other to get the drug ketamine once. Participants will repeat most of the Phase 1 tests.

Phase 3: up to 4 more ketamine doses over 2 weeks.

Participants will have follow-up calls or visits at 6 months and then maybe yearly for 5 years.

DETAILED DESCRIPTION:
A. Objective

Suicide occurs across demographics and psychiatric disorders, killing at least one million individuals worldwide each year. In contrast to other injury-related death such as homicide or motor vehicle accidents, suicide rates have increased, particularly among middle-aged adults. Clinicians have a limited ability to predict imminent suicidal behavior and few, if any, efficacious treatments are available to treat suicidal patients. Advances in the treatment of the suicidal patients have been hampered by an incomplete understanding of the neurobiological underpinnings of the suicidal crisis, as suicidal thoughts and behaviors have not been clearly linked with specific neural circuits.

The aim of this study is to evaluate possible biomarkers of suicidal thoughts and behaviors in individuals currently experiencing a suicidal crisis. In taking a dimensional approach to suicide research, we will be able to study phenomenology across Research Domain Criteria (RDoC) units of analysis, from genes through circuits to self-report and experimental paradigms. Through this approach, we can identify potential neurobiological risk factors for both short and long-term suicide risk. As a secondary aim, we will use ketamine to identify biomarkers of ketamine response in a sample at acute risk for suicide.

B. Study Population

Five participant populations will be recruited into this protocol in order to encompass the continuum of suicide risk. A total of 325 individuals will be enrolled in the study. Participant populations are individuals with the following conditions: 1.) recent suicidal ideation with intent and/or suicide attempt (Group 1- "active crisis", n= 65); 2) a past history of suicide attempt, but no suicidal behavior in the last year (Group 2, n= 65, "attempters"); 3) anxiety or mood symptoms, but no recent or past suicidal thoughts or behavior (Group 3, n= 65); 4) healthy controls with no psychiatric or suicide history (Group 4, n= 65); and lifetime suicidal thoughts with intent (Group 5, n=65, ideators ).

C. Design

The research protocol will occur across three phases: baseline, ketamine response and optional repeated infusions. All participants will first be consented into Phase I, which may last up to seven days. This baseline phase will entail multimodal assessment, using pathophysiological markers (blood draw, lumbar puncture), neuroimaging (fMRI, MEG), polysomnography, clinical ratings and experimental paradigms (shock experiments). Participants will receive their regularly scheduled daily medications, but will not receive additional treatment (including new prn medications, such as benzodiazepines for management of anxiety or agitation) during this brief baseline phase. After completion of Phase I, eligible participants from Group 1 or 5 only (active crisis or ideators) will be offered participation in Phase II, the ketamine response phase. This phase, which will last up to four days, consists of a single, open-label trial of ketamine (0.5 mg/kg). The focus of this phase will be identification of potential biomarkers of antisuicidal ketamine response. Participants who complete Phase II will be offered Phase III, which will involve repeated ketamine infusions over two weeks (2 times/ per week for 2 weeks). Psychiatric medication adjustment will be permitted during Phase III.

After participation in Phases I-III, participants in Groups 1-3 and 5 will be offered standard clinical treatment (excluding healthy controls), or participation in another protocol. In standard clinical treatment, adjustment of psychiatric medications and commencement of psychotherapeutic interventions will be permitted. Finally, participants in Groups 1-3 and 5 will receive follow-up evaluations at six months after completion of Study Phase I.

D. Outcome Measures

In Phase I, the outcome measures will be underlying psychiatric, psychological, neuroimaging, sleep and biological differences between the participant groups. In Phase II, the outcome measures will be reductions in suicidal thoughts and depressive and anxiety symptoms at 24 hours post-ketamine infusion.

ELIGIBILITY:
* INCLUSION CRITERIA:

Phase I: Groups 1-3 and 5 (Patients)

1. 18 to 70 years of age.
2. A level of understanding sufficient to agree to all required tests and examinations, sign an informed consent document and verify understanding by a score >= 90% on the Baseline consent quiz
3. Individuals who are able to get pregnant must be willing to remain sexually abstinent or use at least one form of effective birth control during participation in Phase I.
4. Additional Criteria for Group 1 (Active Crisis): Agree to be hospitalized

Phase I: Group 4 (Healthy Volunteers)

1. 18 to 70 years of age.
2. A level of understanding sufficient to agree to all required tests and examinations, sign an informed consent document.
3. Individuals who are able to get pregnant must be willing to remain sexually abstinent or use at least one form of effective birth control during participation in Phase I.

Phase II: Group 1 (Active Crisis) and Group 5 (Suicide Ideators)

1. Patients must have completed Study Phase I as a participant in Group 1 or 5
2. Participants must verify understanding of the protocol by a score >= 80% on the Ketamine Response consent quiz.
3. Patients in Group 1 or 5 must report at least minimal suicidal ideation, depressive or anxiety symptoms to be eligible for this phase.

   * MADRS score of over 10 (10 used as an outcome measure for remission)126
   * OR HAMA score of over 7 (7 used as an outcome measure for remission)127
   * OR SSI score of 2 or more (indicates any residual suicidal thoughts)
4. Individuals who are able to get pregnant must be willing to remain sexually abstinent or use at least one form of effective birth control during participation in Phase II.

Phase III: Group 1 (Active Crisis) and Group 5 (Suicide Ideators)

1. Participants must have met all inclusion criteria for and completed Study Phase II as a participant in Group 1 (active crisis) or Group 5 (Suicide Ideators).
2. Individuals who are able to get pregnant must be willing to remain sexually abstinent or use at least one form of effective birth control during participation in Phase III.

EXCLUSION CRITERIA:

Phase I: Groups 1-3 and 5 (Patients)

1. Current psychotic features or cognitive impairment that would preclude understanding of the consenting process or tests/examinations.
2. Current drug or alcohol dependence
3. Currently intoxicated or under the acute effects of an illicit substance will not be consented into the study.
4. Pregnant or nursing individuals or those who plan to become pregnant.
5. Serious, unstable medical conditions/problems including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including blood pressure, ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
6. Clinically significant abnormal laboratory tests.
7. Positive HIV test
8. Participants who, in the investigator s judgment, pose a current homicidal risk or pose suicide risk that cannot be managed in a secure, voluntary inpatient setting.
9. Non-English speakers
10. Additional Criteria for Group 1 (Active Crisis): For participants who still experience the effects of their suicide attempt, i.e. someone who overdosed is significantly drowsy or confused, the consenting process will occur after the patient has improved from the effects. If there is a concern around a participant's capacity to consent, the Human Subjects Protections Unit (HSPU) team member who is

monitoring the informed consent process will complete a capacity assessment. Participants who are determined not to have capacity to consent to research will not be included in the study.

Phase I: Group 4 (Healthy Volunteers)

1. Current or past Axis I diagnosis
2. Presence of medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications.
3. Current or past alcohol or substance abuse or dependence diagnosis (except for nicotine or caffeine) (or "substance abuse disorder" per DSM-V).
4. Presence of psychiatric disorders or a history of suicide attempt or death in first-degree relatives.
5. Pregnant or nursing individuals or those who plan to become pregnant.
6. No lifetime suicide attempts or ideations
7. Non-English speakers
8. Positive HIV test

Exclusions for Imaging:

1. Participants with metal objects implanted in the body, such as aneurysm clips, neural stimulators, implanted cardiac pacemakers, or auto-defibrillator, cochlear implant, or ocular foreign body which would make having an MRI scan unsafe
2. Participants who are uncomfortable in small closed spaces (have claustrophobia) and would feel uncomfortable in the MRI machine
3. Participants with a brain abnormality on an initial MRI scan
4. Subjects with hearing loss that has been clinically evaluated and diagnosed and may be worsened through participation in imaging procedures

Phase II: Group 1 (Active Crisis) and Group 5 (Suicide Ideators)

1. Treatment with a reversible MAOI within 2 weeks prior to study Phase II.
2. Treatment with any other concomitant medication not allowed within 5 1/2 half-lives prior to study Phase II.
3. Subjects with one or more seizures without a clear and resolved etiology
4. Participants with a positive urine for an illicit substance no more than 24 hours prior to the ketamine infusion.
5. Presence of current psychotic features or a diagnosis of Schizophrenia or any other psychotic disorder as defined in the DSM-IV or DSM-V
6. Pregnant or nursing individuals or those who plan to become pregnant.
7. A medical finding or condition that in the clinical judgement of the investigator increases the risk of adverse effects from the ketamine administration (for example: findings suggesting difficulties with kidney or cardiac function that may be contraindications for an experimental intervention).

Phase III: Repeated Administration (Group 1) and Group 5 (Suicide Ideators)

1. Intolerable or serious adverse reaction to ketamine during Phase II
2. Treatment with a reversible MAOI within 2 weeks prior to study Phase III.
3. Treatment with any other concomitant medication not allowed within 5 1/2 half-lives prior to study Phase III.
4. Subjects with one or more seizures without a clear and resolved etiology
5. Participants with a positive urine for an illicit substance no more than 24 hours prior to each ketamine infusion.
6. Presence of current psychotic features or a diagnosis of Schizophrenia or any other psychotic disorder as defined in the DSM-IV or DSM-V
7. Pregnant or nursing individuals or those who plan to become pregnant.

Exclusions for Imaging:

1. Participants with metal objects implanted in the body, such as aneurysm clips, neural stimulators, implanted cardiac pacemakers, or auto-defibrillator, cochlear implant, or ocular foreign body which would make having an MRI scan unsafe
2. Participants who are uncomfortable in small closed spaces (have claustrophobia) and would feel uncomfortable in the MRI machine
3. Participants with a brain abnormality on an initial MRI scan
4. Subjects with hearing loss that has been clinically evaluated and diagnosed and may be worsened through participation in imaging procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2030-07-21 (Estimated); Study Completion 2030-07-21 (Estimated)

PRIMARY OUTCOMES:
Study as Whole: Psychiatric, psychological, neuroimaging, sleep and biological differences between participants in Groups 1, 2, 3, 4, and 5 | multiple time-points
  Clinical and research data and samples
Phase II: Scale for Suicide Ideation | multiple time-points
  Clinical rating scale of suicidal ideation
Phase II: Montgomery-Asberg Depression Rating Scale | multiple time-points
  Clinical rating scale of depression
Phase II: Hamilton Psychiatric Rating Scale for Anxiety | multiple time-points
  Clinical rating scale of depression
Phase II: Clinical Global Impression Scale | multiple time-points
  Clinical rating scale of psychiatric symptomology

SECONDARY OUTCOMES:
Anhedonia and Hopelessness via the Snaith-Hamilton Pleasure Scale & the Beck Hopelessness Scale | multiple time-points
  Clinical rating scale of anhedonia and hopelessness
Baseline and Response Biomarkers | multiple time-points
  Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical and demographic and biomarker participant data collected during the trial, after deidentification.
Supporting Information: SAP
Time Frame: Starting within 1 year of completion of the study.
Access Criteria: The Branch Chief will review requests and access will need to be approved by the NIMH/DIRP SD and OCD NIMH and the NIH IRB.

REFERENCES:
- [Derived] Hu H, Lee Y, Tillman AN, Ballard ED, Waldman L, Yuan P, Johnston JN, Peng S, Kvarta MD, Verbalis JG, Zarate CA Jr. Blunted arginine vasopressin secretion in individuals experiencing a major depressive episode with comorbid post-traumatic stress disorder: Results from an exploratory study using copeptin as a surrogate marker. J Neuroendocrinol. 2026 Jan;38(1):e70133. doi: 10.1111/jne.70133. PMID 41555748
- [Derived] Lee Y, Gilbert JR, Waldman LR, Zarate CA Jr, Ballard ED. Potential association between suicide risk, aggression, impulsivity, and the somatosensory system. Soc Cogn Affect Neurosci. 2024 Jul 2;19(1):nsae041. doi: 10.1093/scan/nsae041. PMID 38874947
- [Derived] Lamontagne SJ, Gilbert JR, Zabala PK, Waldman LR, Zarate CA Jr, Ballard ED. Clinical, behavioral, and electrophysiological profiles along a continuum of suicide risk: evidence from an implicit association task. Psychol Med. 2024 May;54(7):1431-1440. doi: 10.1017/S0033291723003331. Epub 2023 Nov 24. PMID 37997749
- [Derived] Ballard ED, Park LT, Pao M, Zarate CA. Clinical Trials With Suicidal Individuals Can Be Conducted Safely. J Clin Psychiatry. 2020 Aug 4;81(5):20l13353. doi: 10.4088/JCP.20l13353. No abstract available. PMID 32757505
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-M-0188.html